CLINICAL TRIAL: NCT07211295
Title: Accurate AI-based Characterisation of Surface Size, Depth and Tissue Composition in Hard-to-Hea Woundsl
Brief Title: Accurate AI-based Characterisation of Surface Size, Depth and Tissue Composition in Hard-to-Heal Wounds
Acronym: SeeWound2
Status: Completed | Type: Observational
Sponsor: University Hospital, Linkoeping (Other)
Responsible Party: Principal Investigator, Folke Sjoberg, Prof, University Hospital, Linkoeping
Other Study IDs: CIP-MDR-SWD001-V1.0-2025, ver,
Record Dates: First submitted 2025-08-31; First posted 2025-10-07 (Actual); Last update posted 2025-10-07 (Actual); Status verified 2025-09

CONDITIONS: Difficult to Heal Wounds
Keywords: VLU; difficult to heal wounds; diabete; ulcers;
MeSH Terms: conditions — Ulcer

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Cohort: cohort

SUMMARY:
This study aims to determine and evaluate the clinical accuracy, precision, and safety of SeeWound 2, an AI-driven wound assessment application, designed for the measurement of wound surface area (cm²), wound depth (mm), and the estimation of the proportion of fibrin covering (slough) and necrosis (%) in real-world clinical settings for patients with hard-to-heal wounds. The study also seeks to validate the non-invasive method for measuring wound depth, as current standard care involves invasive probing of the wound to estimate depth - a practice that this investigational device is intended to replace with a digital, contact-free measurement approach.

DETAILED DESCRIPTION:
SeeWound 2 is a software-based medical device that utilises artificial intelligence to classify and quantify wound tissue types, specifically fibrin covering (slough) and necrosis, as well as to measure wound surface area and depth through digital image analysis. The system operates as a mobile camera-based application, whereby healthcare professionals capture an image of a hard-to-heal wound. The software then automatically analyses the image using integrated AI models in combination with the LiDAR sensor technology embedded in the mobile camera hardware. The product's capability to automatically measure wound surface area, estimate wound depth in a non-invasive manner, and objectively quantify the proportion of slough and necrosis within the wound bed represents a novel functionality not currently available in clinical practice.

ELIGIBILITY:
Inclusion Criteria:

Older than 18 years, men and women Difficult to heal wounds due to diabetes, VLU; Pressure wounds wound larger than 0.5 cm2

Exclusion Criteria:

Exclusion Criteria / Contraindications

Use of SeeWound 2 is not intended for, or is contraindicated in, the following situations:

Patients under 18 years of age. Wounds located in anatomical regions where the full wound surface and depth cannot be captured (e.g. deep fistulas, tunnels, or undermined areas not accessible through surface imaging).

Wounds with excessive exudation or infection that prevents adequate visual assessment.

Patients who are unable or unwilling to provide informed consent. Patients with a known allergy or adverse reaction to any component used in the image acquisition process (where applicable).

Wounds with specific identifiable attributes (e.g. on the face, or containing birthmarks or tattoos) where ethical considerations regarding data handling apply.

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: ntended Use / Target Population The intended target population for SeeWound 2 comprises patients with hard-to-heal wounds. The device is designed for use by qualified healthcare professionals for the clinical assessment, documentation, and monitoring of chronic and complex wounds, including but not limited to venous leg ulcers, diabetic foot ulcers, and pressure ulcers. SeeWound 2 is intended to support clinical decision-making by providing objective, non-invasive measurements of wound surface area and depth, and by enabling the classification and quantification of wound bed tissue composition (slough and necrosis). The product is not intended to replace clinical judgement but to serve as an adjunctive tool to standard wound care practice.
Sampling Method: Probability Sample
Enrollment: 25 (Actual)
Dates: Start 2025-07-01 (Actual); Primary Completion 2025-09-18 (Actual); Study Completion 2025-09-18 (Actual)

PRIMARY OUTCOMES:
Accuracy | During the study
  Regular outcome measures for a Medical Device
Accurac, Precision, Mean absolute Error (MAE); Coefficient of Variation (CV); SD | During the study
  Regular outcome measures for a Medical Device

CONTACTS AND LOCATIONS:
Locations (1):
- BRIVA, Intensive Care for Burns,, Linköping, Östergötland County, Sweden

IPD SHARING:
Plan to Share IPD: No